CLINICAL TRIAL: NCT04022044
Title: Postoperative Changes in Head and Neck Cancer Patients Undergoing Surgery
Status: Completed | Type: Observational
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Other Study IDs: Postoperative changes H&N
Record Dates: First submitted 2019-07-10; First posted 2019-07-16 (Actual); Last update posted 2019-07-16 (Actual); Status verified 2019-07

CONDITIONS: Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Observational group

SUMMARY:
The aim of this study is to evaluate the postoperative changes after a major surgery in head and neck cancer patients. Each participant will be evaluated three times: (1) One day before surgery; (2) one month postoperative and (3) three months postoperative. Assessments included blood pressure, anthropometric measurements, physical measurements and questionnaires on quality of life, nutritional status and cancer symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of head and neck cancer patients planned for an elective major surgery
* More than 18 years of age
* Able to read, write and understand French

Exclusion Criteria:

- Neurological or orthopedic impairments not suitable for testing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with head and neck cancer planned for an elective major surgery
Sampling Method: Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2014-12-30 (Actual); Primary Completion 2019-03-14 (Actual); Study Completion 2019-06-14 (Actual)

PRIMARY OUTCOMES:
Change in functional exercise capacity | Assessments one day before surgery, 1 and 3 months postoperative
  Functional exercise capacity is measured by a 6-minute walk test

SECONDARY OUTCOMES:
Change in muscle fatigability | Assessments one day before surgery, 1 and 3 months postoperative
  Muscle fatigability is measured using a Cybex dynamometer
Change in flexibility | Assessments one day before surgery, 1 and 3 months postoperative
  Flexibility is measured by Toe touch test
Change in flexibility | Assessments one day before surgery, 1 and 3 months postoperative
  Flexibility is measured by sit and reach test
Change in upper body strength and endurance | Assessments one day before surgery, 1 and 3 months postoperative
  Upper body strength and endurance are measured by the 30-second arm curl test
Change in hand grip strength | Assessments one day before surgery, 1 and 3 months postoperative
  Hand grip strength test is performed using a Jamar® dynamometer
Change in health-related quality of life | Assessments one day before surgery, 1 and 3 months postoperative
  Health-related quality of life is evaluated with the version 4 of the University of Washington head and neck cancer questionnaire
Change in common symptom batteries in cancer patients | Assessments one day before surgery, 1 and 3 months postoperative
  Common symptom batteries is measured by the Edmonton Symptom Assessment System (revised version) questionnaire
Change in nutritional status | Assessments one day before surgery, 1 and 3 months postoperative
  Nutritional status is measured with the Short Nutritional Assessment Questionnaire
Change in blood pressure | Assessments one day before surgery, 1 and 3 months postoperative
  Resting blood pressure is measured using the M6 Comfort automatic blood pressure monitor
Change in weight | Assessments one day before surgery, 1 and 3 months postoperative
  Weight (kg) is measured by using a bioelectrical impedance analysis
Change in fat body mass | Assessments one day before surgery, 1 and 3 months postoperative
  Fat body mass (%) is measured by using a bioelectrical impedance analysis
Change in waist circumference | Assessments one day before surgery, 1 and 3 months postoperative
  Waist circumference is measured with a non-elastic tape measure

IPD SHARING:
Plan to Share IPD: Undecided